CLINICAL TRIAL: NCT03451201
Title: Effect of High-Intensity Interval Exercise Training Compared With Moderate-intensity Continuous Training on Endothelial Function and Cardiorespiratory Fitness of Type 1 Diabetes Patients
Brief Title: High-Intensity Exercise and Endothelial Function in Type 1 Diabetes(HIIT-T1D)
Acronym: HIIT-T1D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 150564
Record Dates: First submitted 2018-02-23; First posted 2018-03-01 (Actual); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Type 1 Diabetes Mellitus; Endothelial Dysfunction
Keywords: Exercise; High-Intensity Interval Training; Type 1 diabetes; Endothelial Dysfunction
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Randomised Clinical Trial, 3 parallel groups: HIIT ( High-Intensity Interval Training) MCT (moderate intensity continuous training) and Sedentary Control Group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High Intensity Interval Training (Experimental): High Intensity Interval Exercise Training in cycle ergometer 3 times a week for 8 weeks
  Interventions: Behavioral: High Intensity Interval Training
- Moderate Continuous Exercise Training (Active Comparator): Moderate Continuous Interval Training
  Interventions: Behavioral: Moderate Continuous Exercise Training
- Non-exercise (Other): Sedentary Type 1 Diabetes Controls.
  Interventions: Other: Non-exercise

INTERVENTIONS:
Behavioral: High Intensity Interval Training — High Intensity Interval Exercise Training in cycle ergometer, exercising at 80% of maximal capacity during one minute alternated with exercise at 50% of maximal capacity during 4 minutes intervals, for a total of 30 minutes. Three times a week for 8 weeks
  Arms: High Intensity Interval Training
Behavioral: Moderate Continuous Exercise Training — Moderate Continuous Exercise Training 3 times a week for 8 weeks at 50% of maximal capacity
  Arms: Moderate Continuous Exercise Training
Other: Non-exercise — Conventional care for sedentary Type 1 Diabetes Controls. No intervention.
  Arms: Non-exercise

SUMMARY:
To study the effect of 8 week high-intensity interval training (HIIT) compared with moderate intensity (MCT) interval training and sedentary patients(CON) with type 1 diabetes. Adult T1DM patients without known complications are randomised in blocks into these 3 groups according to their baseline flow mediated dilation (FMD). After 8 week exercise training, the main outcome, FMD, is re-evaluated. Additional variables such as VO2 peak for cardiovascular fitness, oxidative stress and endothelial independent vasodilation to study vascular rigidity are also evaluated.

DETAILED DESCRIPTION:
In a randomized controlled open trial, 36 adult type 1 diabetes mellitus (T1DM) patients without known complications were randomized into 3 groups: HIIT n=12; MCT n=12 and a sedentary control group (CON) n=12. Total sample size was calculated to a power of 80% alha 0.05 and a difference in mean FMD of 2%. Before randomisation, flow mediated dilation (FMD) and maximal exercise capacity (VO2 peak)is determined. Block Randomisation based on FMD rank values are done to equalize baseline FMD. Exercise sessions are performed in cycle ergometers during 40 minutes, 3 times a week, along 8 weeks. HIIT protocol, intensity vary from 50 to 85% of the maximum heart rate (HRmax), while in MCT, HR remained stable at 50% HRmax. Endothelial function was measured by flow mediated dilation (FMD) for endothelium-dependent vasodilation (EDVD) and smooth-muscle function was measured by nitroglycerine mediated dilation (endothelium independent vascular dilation) - (EIVD). Peak oxygen consumption (VO2peak) and oxidative stress markers were determined before and after the training period. ED was defined as an increase of less than 8% in vascular diameter after cuff release.

ELIGIBILITY:
Inclusion Criteria:

T1DM

* Physically inactive or not involved in exercise training programs in the previous 6 months
* Interested in starting an exercise training program.

Exclusion Criteria:

* Smokers,
* Pregnancy
* Co-morbidities not related to diabetes
* Drugs other than insulin
* Loss of renal function (serum creatinine above 1.5 mg/dl),
* Moderate to severe retinopathy or blindness,
* Suspected or confirmed coronary artery disease,
* Severe peripheral neuropathy
* Foot ulcers or history of previous foot ulcer
* Suspected or confirmed clinical autonomic neuropathy.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Endothelial Dependent Mediated Vascular Dilation | 8 weeks
  Percent of change from baseline in flow mediated dilation measured through arterial ultrasound at right arm

SECONDARY OUTCOMES:
Peak oxygen consumption | 8 weeks
  Percent of change in maximal oxygen capacity measured by in maximal oxygen consumption
Endothelial independent vascular dilation | 8 weeks
  Percent of change from baseline in nitrate mediated dilation measured through arterial ultrasound at right arm

CONTACTS AND LOCATIONS:
Overall Officials: Marcello C Bertoluci, MD, PhD, Principal Investigator — Hospital de Clinicas de Porto Alegre
Locations (1):
- Serviço de Endocrinologia e Metabologia do HCPA, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mitranun W, Deerochanawong C, Tanaka H, Suksom D. Continuous vs interval training on glycemic control and macro- and microvascular reactivity in type 2 diabetic patients. Scand J Med Sci Sports. 2014 Apr;24(2):e69-76. doi: 10.1111/sms.12112. Epub 2013 Sep 17. PMID 24102912
- [Background] Corretti MC, Anderson TJ, Benjamin EJ, Celermajer D, Charbonneau F, Creager MA, Deanfield J, Drexler H, Gerhard-Herman M, Herrington D, Vallance P, Vita J, Vogel R; International Brachial Artery Reactivity Task Force. Guidelines for the ultrasound assessment of endothelial-dependent flow-mediated vasodilation of the brachial artery: a report of the International Brachial Artery Reactivity Task Force. J Am Coll Cardiol. 2002 Jan 16;39(2):257-65. doi: 10.1016/s0735-1097(01)01746-6. PMID 11788217
- [Background] Ce GV, Rohde LE, da Silva AM, Punales MK, de Castro AC, Bertoluci MC. Endothelial dysfunction is related to poor glycemic control in adolescents with type 1 diabetes under 5 years of disease: evidence of metabolic memory. J Clin Endocrinol Metab. 2011 May;96(5):1493-9. doi: 10.1210/jc.2010-2363. Epub 2011 Feb 23. PMID 21346068
- [Background] Bertoluci MC, Ce GV, da Silva AM, Wainstein MV, Boff W, Punales M. Endothelial dysfunction as a predictor of cardiovascular disease in type 1 diabetes. World J Diabetes. 2015 Jun 10;6(5):679-92. doi: 10.4239/wjd.v6.i5.679. PMID 26069717
- [Background] Seeger JP, Thijssen DH, Noordam K, Cranen ME, Hopman MT, Nijhuis-van der Sanden MW. Exercise training improves physical fitness and vascular function in children with type 1 diabetes. Diabetes Obes Metab. 2011 Apr;13(4):382-4. doi: 10.1111/j.1463-1326.2011.01361.x. PMID 21226819
- [Background] Molmen-Hansen HE, Stolen T, Tjonna AE, Aamot IL, Ekeberg IS, Tyldum GA, Wisloff U, Ingul CB, Stoylen A. Aerobic interval training reduces blood pressure and improves myocardial function in hypertensive patients. Eur J Prev Cardiol. 2012 Apr;19(2):151-60. doi: 10.1177/1741826711400512. Epub 2011 Mar 4. PMID 21450580
- [Derived] Eckstein ML, Farinha JB, McCarthy O, West DJ, Yardley JE, Bally L, Zueger T, Stettler C, Boff W, Reischak-Oliveira A, Riddell MC, Zaharieva DP, Pieber TR, Muller A, Birnbaumer P, Aziz F, Brugnara L, Haahr H, Zijlstra E, Heise T, Sourij H, Roden M, Hofmann P, Bracken RM, Pesta D, Moser O. Differences in Physiological Responses to Cardiopulmonary Exercise Testing in Adults With and Without Type 1 Diabetes: A Pooled Analysis. Diabetes Care. 2021 Jan;44(1):240-247. doi: 10.2337/dc20-1496. Epub 2020 Nov 12. PMID 33184152
- [Derived] Boff W, da Silva AM, Farinha JB, Rodrigues-Krause J, Reischak-Oliveira A, Tschiedel B, Punales M, Bertoluci MC. Superior Effects of High-Intensity Interval vs. Moderate-Intensity Continuous Training on Endothelial Function and Cardiorespiratory Fitness in Patients With Type 1 Diabetes: A Randomized Controlled Trial. Front Physiol. 2019 Apr 24;10:450. doi: 10.3389/fphys.2019.00450. eCollection 2019. PMID 31110479